CLINICAL TRIAL: NCT00478049
Title: A Randomized, Open Label, Parallel Group, Regional, Multicenter, Phase III Study of Oral Gefitinib (IRESSA®) Versus Intravenous Docetaxel (TAXOTERE®) in Patients With Locally Advanced or Metastatic Recurrent Non Small Cell Lung Cancer Who Have Previously Received Platinum Based Chemotherapy (ISTANA)
Brief Title: Iressa as Second Line Therapy in Advanced NSCLC-Asia
Acronym: ISTANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7913L00039
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: NSCLC
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel

ARMS (2):
- 1 (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel
- 2 (Experimental): Gefitinib
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg oral tablet
  Other Names: ZD1839; IRESSA
  Arms: 2
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere
  Arms: 1

SUMMARY:
This is a randomized, open-label, parallel group, phase III, multicenter, regional study. The total number of patients expected to be exposed to study procedures is approximately 150 patients will be recruited by investigational sites throughout the Asia Pacific region that have expertise in treating patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell bronchogenic carcinoma: adenocarcinoma (including bronchoalveolar), squamous cell carcinoma, large cell carcinoma or mixed (adenocarcinoma and squamous) or undifferentiated carcinoma.
* WHO Performance status 0-2
* NSCLC - locally advanced (Stage IIIB) or metastatic (stage IV) disease, not amenable to curative surgery or radiotherapy
* Life expectancy of 12 weeks.

Exclusion Criteria:

* ALT/AST: >2.5x ULRR if no demonstrable liver metastases or greater than 5 x ULRR in the presence of liver.
* Inadequate bone marrow function; Absolute neutrophil count: <1.5 x 109/L, Platelets: < 100 x 109/L
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma of skin or cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Compare progression free survival between patients on gefitinib or on docetaxel by Progression as per Response Evaluation Criteria In Solid Tumors | Survival

SECONDARY OUTCOMES:
To compare the overall objective tumor response rates between patients on gefitinib or on docetaxel by overall objective tumor response (complete response (CR) + partial response (PR)) using RECIST criteria. | Survival
To compare changes in quality of life (QoL) between patients on gefitinib or on docetaxel by QoL as measured by the FACT-L total score | Every Visit
For those patients who are symptomatic at baseline to compare improvement in symptom control between patients on gefitinib or on docetaxel by the FACT-L LCS (Functional Assessment of Cancer Therapy - Lung Lung Cancer Subscale). | Each Visit
To compare the safety and tolerability of gefitinib and of docetaxel by Frequency and severity of adverse events (AEs) and laboratory parameters. | Every Visit

CONTACTS AND LOCATIONS:
Overall Officials: SangWe Kim, MD, Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Research Site, Incheon
  - Research Site, Kyonggi-do
  - Research Site, Seoul
  - Research Site, Suwon